CLINICAL TRIAL: NCT00214578
Title: Seroquel on Glucose Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1441C00125
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Seroquel (quetiapine)

SUMMARY:
The purpose of this study is to determine whether six months treatment with the antipsychotic medicine Seroquel (quetiapine) may affect the schizophrenic patient's glucose metabolism

ELIGIBILITY:
Inclusion Criteria:

* In- or outpatients with schizophrenia, 18-65 years old, requiring a change in treatment due to insufficient efficacy or tolerability and giving signed informed consent.

Exclusion Criteria:

* Known diabetes mellitus, high HbA1c, fasting plasma glucose and/or high 2h glucose-OGTT.
* Previous use of atypicals (3 months) or other medications that might influence glucose metabolism
* Contraindications or non-responsiveness for any of the treatments or other safety issues
* Expected non-compliance to treatment and/or study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572
Dates: Start 2004-04; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To analyze the safety/tolerability profile of quetiapine on glucose metabolism in schizophrenic patients

SECONDARY OUTCOMES:
Glucose metabolism, blood lipid levels and weight

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca CNS Medical Group, Study Director — AstraZeneca
Locations (70):
- Bulgaria (5):
  - Research Site, Burgas
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Sofia- Novi Iskar
  - Research Site, Varna
- Czechia (8):
  - Research Site, Dobjany
  - Research Site, Dob¿any U Plzn¿
  - Research Site, Havlí¿k¿v Brod
  - Research Site, Kladno
  - Research Site, Miro¿ov
  - Research Site, Opava
  - Research Site, Pilsen
  - Research Site, Prague
- Germany (13):
  - Research Site, Tübingen, Baden-Wurttemberg
  - Research Site, München, Bavaria
  - Research Site, Bonn, North Rhine-Westphalia
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Herten
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Tübingen
- Hungary (10):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gy¿r
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Szeged
  - Research Site, Szolnok
- Norway (7):
  - Research Site, Bergen
  - Research Site, Drammen
  - Research Site, Hagavik
  - Research Site, Stavanger
  - Research Site, Stokmarknes
  - Research Site, Straume
  - Research Site, Tønsberg
- Romania (3):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Iași
- Slovakia (12):
  - Research Site, Banská Bystrica
  - Research Site, Bojnice
  - Research Site, Bratislava
  - Research Site, Domaša
  - Research Site, Ko¿ice
  - Research Site, Liptovský Mikulá¿
  - Research Site, Michalovce Strá¿any
  - Research Site, Nitra
  - Research Site, Pre¿ov
  - Research Site, Rimavská Sobota
  - Research Site, ¿ilina-Byt¿ica
  - Research Site, ¿ilina
- South Africa (10):
  - Research Site, Medunsa, Pretoria
  - Research Site, Bloemfontein
  - Research Site, CapeTown
  - Research Site, Durban
  - Research Site, Ga-Rankuwa
  - Research Site, Johannesburg
  - Research Site, Krugersdorp
  - Research Site, Parktown
  - Research Site, Pretoria
  - Research Site, Tygerberg
- United Kingdom (2):
  - Research Site, Sutton Coldfield, West Midlands
  - Research Site, Birmingham

REFERENCES:
- [Derived] Newcomer JW, Ratner RE, Eriksson JW, Emsley R, Meulien D, Miller F, Leonova-Edlund J, Leong RW, Brecher M. A 24-week, multicenter, open-label, randomized study to compare changes in glucose metabolism in patients with schizophrenia receiving treatment with olanzapine, quetiapine, or risperidone. J Clin Psychiatry. 2009 Apr;70(4):487-99. doi: 10.4088/jcp.08m04132. Epub 2009 Apr 7. PMID 19358783